CLINICAL TRIAL: NCT01603641
Title: BOTOX® Treatment in Pediatric Lower Limb Spasticity: Open-label Study
Brief Title: BOTOX® Open-Label Treatment in Pediatric Lower Limb Spasticity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191622-112; 2012-000084-24 (EudraCT Number)
Record Dates: First submitted 2012-05-21; First posted 2012-05-22 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-07

CONDITIONS: Pediatrics; Muscle Spasticity; Cerebral Palsy
MeSH Terms: conditions — Muscle Spasticity; Cerebral Palsy | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BOTOX® (Experimental): Participants received maximum of 5 treatments of intramuscular injections of BOTOX® (botulinum toxin Type A) into a single lower limb muscles or divided between both lower limb muscles or into the lower limb muscles and/or upper limb muscles at a minimum of 12 weeks apart. Treatment dosing was according to investigator judgment not to exceed a maximum of 8 unit per kilogram (U/kg) of body weight (not to exceed 300 U) in treatment Cycle 1. Dose could be increased to a maximum of 10 U/kg (not to exceed 340 U) in treatment Cycles 2-5. Participants received intramuscular injections of BOTOX® (botulinum toxin Type A) 4 or 8 U/kg into the lower limb in the previous study or were de novo participants who were not enrolled in the previous study.
  Interventions: Biological: Botulinum Toxin Type A

INTERVENTIONS:
Biological: Botulinum Toxin Type A — Participants received intramuscular injections of botulinum toxin Type A into the lower limb muscles and/or upper limb muscles at a minimum of 12 weeks apart for a maximum of 5 treatments.
  Other Names: BOTOX®; OnabotulinumtoxinA

SUMMARY:
This study will evaluate the long-term safety of BOTOX® (botulinum toxin Type A) for the treatment of pediatric lower limb spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Minimum weight of 10 kilograms (kg)/22 pounds (lb)
* Cerebral palsy with dynamic muscle contracture of the ankle

Exclusion Criteria:

* Muscular dystrophy, myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or mitochondrial disease
* Uncontrolled epilepsy
* Botulinum Toxin therapy of any serotype for any condition within the last 3 months
* History of surgical intervention of the lower study leg within 1 year, or planned surgery of any limb during the study

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 370 (Actual)
Dates: Start 2012-11-05 (Actual); Primary Completion 2018-08-25 (Actual); Study Completion 2018-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily McCusker, Study Director — Allergan
Locations (56):
- United States (26):
  - ABS Health, LLC, Pasadena, California
  - Harrison Clinical Management, Pomona, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Associated Neurologists of Southern Connecticut, P.C., Fairfield, Connecticut
  - New England Institute for Clinical Research, Stamford, Connecticut
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Axcess Medical Research, LLC, Loxahatchee Groves, Florida
  - Pediatric Neurology, P.A., Orlando, Florida
  - Children's Healthcare of Atlanta Children's Rehabilitation Associates, Atlanta, Georgia
  - Shirley Ryan Ability Lab, Chicago, Illinois
  - Beaumont Children's Hospital Pediatric Research, Royal Oak, Michigan
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Clinical Research Center of New Jersey, Voorhees Township, New Jersey
  - NYU Hospital for Joint Diseases, New York, New York
  - Columbia University Dept. of Rehab. & Regenerative Medicine, New York, New York
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine Texas Children's Hospital, Houston, Texas
  - Road Runner Research, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
- Hungary (2):
  - Semmelweis Egyetem- Ortopédiai Klinika Karolina út 27, Budapest
  - Debrecen University Clinical Center, Orthopedic Clinic, Debrecen
- Istituto IRCCS G. Salini, Genoa, Italy
- Philippines (3):
  - Philippine Orthopedic Center, Quezon City
  - St. Luke's Medical Center, Quezon City
  - Philippine Children's Medical Center, Quezon City
- Poland (10):
  - Uniwersytecki Dzieciecy Szpita, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Rehabilitacji Krok po Kroku, Gdansk
  - Specjalistyczny Gabinet Neurologiczny, Krakow
  - Centrum Medyczne "POMOC", Lodz
  - INTERMED, Lublin, Lublin
  - CRH ŻAGIEL MED, Lublin, Lublin
  - Szpital Wojewodzki Nr 2, Rzeszów
  - Poradnia Rehab - Neurologiczneij dla Dzieci I Mlodziezy Aga, Warsaw
  - NZOZ Mazowieckie Centrum, Warsaw
- Russia (3):
  - Childrens Republic Hospital, Kazan'
  - Smolensk Regional Hospital- Regional Budget State Healthcare institution, Smolensk
  - Tyumen Regional Hospital #2 - State Budget Healthcare Institution of Tyumen region, Tyumen
- South Korea (6):
  - Daegu Fatima Hospital, Daegu
  - National Health Insurance Service Ilsan Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Thailand (2):
  - Maharaj Nakorn ChiangMai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
- Turkey (Türkiye) (3):
  - Ankara Diskapi Yildrim Beyazit, Ankara
  - Kocaeli Üniversitesi, Kocaeli
  - Selçuk Üniversitesi, Konya

REFERENCES:
- See also: More information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pediatric participants with lower limb spasticity who were previously treated with BOTOX® in study 191622-111 [NCT01603628] and de novo participants received up to 5 BOTOX® treatments in this study.
Period: Overall Study
Arm/Group | BOTOX®
Started | 370
Safety Population (Treated) | 367
Modified Intent-to-treat Population | 366
Completed | 335
Not Completed | 35
Not completed — Did not Receive Treatment | 3
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 6
Not completed — Personal Reasons | 18
Not completed — Other Miscellaneous Reasons | 6

BASELINE CHARACTERISTICS:
Population: Safety population included all treated participants.
Arm/Group | BOTOX®
Number analyzed (Participants) | 367
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.9 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167
  Male | 200
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 224
  Black | 9
  Asian | 109
  Hispanic | 21
  Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. A TEAE was an AE that occurred after receiving the first dose of investigational product or an AE present prior to first dose but increased in severity during the Treatment Period.
Time Frame: From first dose of study drug up to 12 weeks post last dose (Up to 60 weeks)
Population: Safety population included all treated participants.
Measure: Number; unit: percentage of participants
Arm/Group | BOTOX®
Number analyzed (Participants) | 367
percentage of participants | 65.4

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 12 weeks post last dose (Up to 60 weeks)
Description: Safety Population included all treated participants.
Arm/Group | BOTOX®
All-Cause Mortality (participants affected / at risk) | 0/367
Serious Adverse Events (participants affected / at risk) | 24/367
Other Adverse Events (participants affected / at risk) | 145/367
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® (N=367)
Arrhythmia (Cardiac disorders) | 1
Entropion (Eye disorders) | 1
Strabismus (Eye disorders) | 1
Cataract (Eye disorders) | 1
Pharyngitis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 4
Laryngitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Febrile convulsion (Nervous system disorders) | 4
Hemiplegia (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 2
Status epilepticus (Nervous system disorders) | 2
Epilepsy (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® (N=367)
Pyrexia (General disorders) | 27
Upper respiratory tract infection (Infections and infestations) | 67
Nasopharyngitis (Infections and infestations) | 65
Bronchitis (Infections and infestations) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2014-01-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT01603641/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT01603641/SAP_001.pdf